CLINICAL TRIAL: NCT03570476
Title: Open-Label, Pilot Study of Olaparib as a Neoadjuvant Therapy for Patients Undergoing Prostatectomy for Localized Prostate Cancer
Brief Title: Olaparib Before Surgery in Treating Participants With Localized Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to slow accrual
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9985; NCI-2018-00977 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9985 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH); RG1718008 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2018-06-05; First posted 2018-06-27 (Actual); Results first posted 2020-09-21 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-07

CONDITIONS: Prostate Adenocarcinoma Without Neuroendocrine Differentiation; Stage I Prostate Cancer AJCC v8; Stage II Prostate Cancer AJCC v8; Stage IIA Prostate Cancer AJCC v8; Stage IIB Prostate Cancer AJCC v8; Stage IIC Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — olaparib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (olaparib, radical prostatectomy) (Experimental): Participants receive olaparib orally twice daily for 90 days in the absence of unacceptable toxicity. Beginning 1 day after last olaparib dose, participants undergo radical prostatectomy.
  Interventions: Drug: Olaparib; Procedure: Radical Prostatectomy

INTERVENTIONS:
Drug: Olaparib — Given orally
  Other Names: AZD2281; KU-0059436; Lynparza; PARP Inhibitor AZD2281
Procedure: Radical Prostatectomy — Undergo surgery
  Other Names: Prostatovesiculectomy

SUMMARY:
This phase II trial studies how well olaparib works in treating participants with prostate cancer that has not spread to other parts of the body (localized). Olaparib may stop the growth of tumor cells by interfering with the activity of a substance called PARP, which is inside cells. Giving olaparib before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the pathological complete response rate following olaparib when administered as neoadjuvant therapy prior to prostatectomy in patients with localized prostate cancer containing homozygous or complementary deoxyribonucleic acid [DNA] repair deficiency.

SECONDARY OBJECTIVE:

I. To determine the rate of positive surgical margins, extracapsular extension, positive seminal vesicles and lymph nodes at the time of prostatectomy.

OUTLINE:

Participants receive olaparib orally twice daily for 90 days in the absence of unacceptable toxicity. Beginning 1 day after last olaparib dose, participants undergo radical prostatectomy.

After completion of study treatment, participants are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures.
* Histologically confirmed adenocarcinoma of the prostate without morphologic neuroendocrine differentiation or small cell features.
* The presence of homologous recombination deficiency defined by either; A) Inherited pathogenic variant of BRCA2, ATM, BRCA1, PALB2 by a Clinical Laboratory Improvement Act (CLIA) level germline assay or B) have evidence by somatic sequencing using a CLIA level assay of biallelic inactivation of BRCA1, BRCA2, PALB2, FANCA or biallelic inactivation or monoallelic inactivating mutation of ATM. It is anticipated that the majority of patients will be germline carriers of a pathogenic variant of BRCA1, BRCA2 or ATM. Other germline mutations will be considered at investigator's discretion.
* Must be candidates for radical prostatectomy and considered surgically resectable by urologic evaluation.
* No evidence of metastatic disease or nodal disease as determined by radionuclide bone scans and computed tomography (CT)/magnetic resonance imaging (MRI); non-pathological lymph nodes must be less than 20 mm in the short (transverse) axis.
* Provided written authorization for use and release of health and research study information.
* Hemoglobin >= 10.0 g/dL with no blood transfusion in the past 28 days.
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L (within 28 days prior to administration of study treatment).
* Platelet count >= 100 x 10^9/L (within 28 days prior to administration of study treatment).
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (within 28 days prior to administration of study treatment).
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) / alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal unless liver metastases are present in which case they must be =< 5 x ULN (within 28 days prior to administration of study treatment).
* Patients must have creatinine clearance estimated using the Cockcroft-Gault equation of >= 51 mL/min (within 28 days prior to administration of study treatment).
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Patients must have a life expectancy >= 16 weeks.
* Male patients and their partners, who are sexually active and of childbearing potential, must agree to the use of two highly effective forms of contraception in combination throughout the period of taking study treatment and for 3 months after last dose of study drug(s) to prevent pregnancy in a partner.
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
* Any previous treatment with PARP inhibitor, including olaparib.
* Other malignancy within the last 5 years except: adequately treated non-melanoma skin cancer, or other solid tumors including lymphomas (without bone marrow involvement) curatively treated with no evidence of disease for >= 5 years.
* Resting electrocardiogram (ECG) with corrected QT interval (QTc) > 470 msec on 2 or more time points within a 24-hour period or family history of long QT syndrome.
* Patients receiving any systemic chemotherapy, hormonal therapy or radiotherapy.
* Concomitant use of known strong CYP3A inhibitors (e.g. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (e.g. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is 2 weeks.
* Concomitant use of known strong (e.g. phenobarbital, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's wort) or moderate CYP3A inducers (e.g. bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib is 5 weeks for phenobarbital and 3 weeks for other agents.
* Patients with myelodysplastic syndrome/acute myeloid leukemia or with features suggestive of myelodysplastic syndromes (MDS)/acute myeloid leukemia (AML).
* Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery.
* Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, extensive interstitial bilateral lung disease on high resolution computed tomography (HRCT) scan or any psychiatric disorder that prohibits obtaining informed consent.
* Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
* Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV).
* Patients with a known hypersensitivity to olaparib or any of the excipients of the product.
* Patients with known active hepatitis (i.e., hepatitis B or C) due to risk of transmitting the infection through blood or other body fluids.
* Previous allogenic bone marrow transplant or cord blood transplantation.
* Whole blood transfusions in the last 120 days prior to entry to the study (packed red blood cells and platelet transfusions are acceptable).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-09-11 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Montgomery, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Olaparib, Radical Prostatectomy): Participants receive olaparib orally twice daily for 90 days in the absence of unacceptable toxicity. Beginning 1 day after last olaparib dose, participants undergo radical prostatectomy.
  Olaparib: Given PO
  Radical Prostatectomy: Undergo surgery
Period: Overall Study
Arm/Group | Treatment (Olaparib, Radical Prostatectomy)
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment (Olaparib, Radical Prostatectomy): Participants receive olaparib PO BID for 90 days in the absence of unacceptable toxicity. Beginning 1 day after last olaparib dose, participants undergo radical prostatectomy.
  Olaparib: Given PO
  Radical Prostatectomy: Undergo surgery
Arm/Group | Treatment (Olaparib, Radical Prostatectomy)
Number analyzed (Participants) | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response (pCR) Rate
Description: Percent of patients who achieve a pCR at the time of prostatectomy, after 12 weeks of neoadjuvant therapy with olaparib. PCR is defined as the absence of morphologically identifiable carcinoma in the prostatectomy specimen. Assessment will be based on the recommendations of the International Society of Urological Pathology (ISUP).
Time Frame: At time of prostatectomy (at 12 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Olaparib, Radical Prostatectomy)
Number analyzed (Participants) | 2
Participants | 0

2. Primary Outcome: Number of Participants With Adverse Events
Description: Will be evaluated according to Common Terminology Criteria for Adverse Events (CTCAE).
Time Frame: Up to 30 days after the last dose of olaparib
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Olaparib, Radical Prostatectomy)
Number analyzed (Participants) | 2
Participants | 0

3. Secondary Outcome: Rate of Positive Surgical Margins
Description: The rate of detectable tumor in pathology specimens obtained at prostatectomy.
Time Frame: At time of prostatectomy (at 12 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Olaparib, Radical Prostatectomy)
Number analyzed (Participants) | 2
Participants | 0

4. Secondary Outcome: Stage of Disease
Description: Pathology specimens obtained at prostatectomy will be assessed using the tumor, lymph node, and metastasis (TNM) staging system for prostate cancer.
  Stage Stage 2 represents patients with disease without evidence of extension outside of the prostate Stage 3 represents patients with disease which has penetrated the capsule of the prostate
Time Frame: At time of prostatectomy (at 12 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Olaparib, Radical Prostatectomy)
Number analyzed (Participants) | 2
Participants
  Stage 2 | 0
  Stage 3 | 2

ADVERSE EVENTS:
Time Frame: 4 months
Description: Adverse events were collected according to CTCAE version 5
Arm/Group | Treatment (Olaparib, Radical Prostatectomy)
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2019-01-14): https://cdn.clinicaltrials.gov/large-docs/76/NCT03570476/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2020-04-23): https://cdn.clinicaltrials.gov/large-docs/76/NCT03570476/Prot_SAP_001.pdf